# The Impact of the Attention Training Technique on Attention Control and High Worry Study Protocol and Statistical Analysis Plan

NCT03216382

June 10, 2021

### Study Protocol and Statistical Analysis Plan

#### NCT03216382

#### **Protocol**

- Phone screen to assess eligibility
- Visit 1: Baseline
  - Participants completed consent form, a demographic questionnaire, the GAD-Q-IV, MCQ-30, ACS, PSWQ-PW, SMQ, and the CESD-R.
  - o Participants completed the dot-probe task, ANT, and breathing focus task.
  - Participants assigned to complete daily diary every evening, monitoring worry and attention.
- Week 1: Diary
  - o Monitoring worry and attention at home every evening
- Visit 2: Preintervention (1 week after baseline)
  - o Participants completed the MCQ-30, the ACS, the SMQ, and the PSWQ-PW.
  - o Participants completed the dot-probe, ANT, and breathing focus task.
  - Participants randomly assigned to one of the two conditions: attention training or control.
  - o Participants completed self-focused attention rating scale.

- o Participants given rationale (same for both conditions).
- o Participants listened to ATT or control recording.
- Participants recomplete the self-focused attention rating scale and the credibility and expectancy questionnaire.
- Participants asked to listen to assigned recording once per day over the follow week while continuing to monitor worry and attention.

## • Week 2: Recording and Diary

- Participants listened to assigned recording once per day and complete diary every evening.
- Before and after recording, participants completed self-focused attention rating scale. Participants also asked at the end of listening to the recording to what percentage they focused on the recording.
- Visit 3: Postintervention (1 week after preintervention)
  - o Participants completed the MCQ-30, the ACS, and the PSWQ-PW.
  - o Participants completed the dot-probe, the ANT, and the breathing focus task.
  - Participants were debriefed about the goals and hypotheses of the study.
  - Those in the control condition were offered the opportunity to listen to the ATT recording in the lab.

#### **Data Analysis Plan**

Scores from the questionnaires, the ANT, dot-probe task, and breathing focus task were analyzed using a 3x2 repeated measures Oneway Analysis of Variance (ANOVA), with time as a

variable with three levels (visits 1, 2 and 3) and condition as a variable with two levels (ATT and Control). This was a pre-planned analysis.

Diary data were analyzed using hierarchical linear modelling. The proposed structure of the data included 2 levels, the first level representing the data across time points (i.e., an individual's responses over the course of the study), and the second level representing the participant's assigned condition (ATT vs. Control). A piecewise analysis of the data was conducted with a random intercept and fixed slopes. Linear multilevel models were run separately for each outcome variable. Predictor variables included condition, time (piece 1: baseline, or visit 1 to visit 2 and piece 2: intervention period, or visit 2 to visit 3), and an interaction between condition and time. Quadratic models were also run, in case change was not linear. This was a pre-planned analysis.

Only uncontrollability of worry and self-focused attention were analyzed. It was decided post-hoc that uncontrollability and intensity may be redundant, and thus uncontrollability was chosen due to perceived uncontrollability of worry being part of the diagnostic criteria of GAD. Further, minutes of worry and frequency of worry episodes were difficult to interpret, as there was huge variability in responses. Many participants reported that they found it very difficult to quantify their worry in this way and they were not confident in their responses.